CLINICAL TRIAL: NCT00151996
Title: A Phase II, Open-Label Co-Administration Study of SPD503 and Psychostimulants in Children and Adolescents Aged 6-17 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Safety and Tolerability of SPD503 and Psychostimulants in Children and Adolescents Aged 6-17 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD503-205
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Guanfacine; Amphetamine

ARMS (2):
- Methylphenidate + SPD503 (Experimental)
  Interventions: Drug: Methylphenidate + SPD503 (Guanfacine hydrochloride)
- Amphetamine + SPD503 (Experimental)
  Interventions: Drug: Amphetamine + SPD503

INTERVENTIONS:
Drug: Methylphenidate + SPD503 (Guanfacine hydrochloride)
  Arms: Methylphenidate + SPD503
Drug: Amphetamine + SPD503
  Arms: Amphetamine + SPD503

SUMMARY:
The purpose of this study is to assess the safety and tolerability of administering SPD503 (Guanfacine hydrochloride) with psychostimulants (amphetamine or methylphenidate) for treatment of ADHD in children and adolescents aged 6-17

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a primary diagnosis of ADHD
* Subject on a stable dose of a psychostimulant approved for the treatment of ADHD for at least 1 month, with sub-optimal control in the Investigator's opinion
* Male or non-pregnant female subject who agrees to comply with any applicable contraceptive requirements

Exclusion Criteria:

* Subject has current uncontrolled comorbid psychiatric diagnosis (except ODD and mild anxiety) with significant symptoms
* History of seizure during the last 2 years
* Subject has any specific cardiac condition or family history of significant cardiac condition
* Subject is pregnant or lactating

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2004-08-16 (Actual); Primary Completion 2004-12-27 (Actual); Study Completion 2004-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Result] Spencer TJ, Greenbaum M, Ginsberg LD, Murphy WR. Safety and effectiveness of coadministration of guanfacine extended release and psychostimulants in children and adolescents with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2009 Oct;19(5):501-10. doi: 10.1089/cap.2008.0152. PMID 19877974
- See also: FDA-approved label — http://www.intuniv.com/documents/INTUNIV_Full_Prescribing_Information.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Dose titration of SPD503 (Guanfacine HCl) for 3 weeks starting at 1 mg/day and increased in 1 mg weekly increments up to 4 mg/day (or to the highest tolerated dose); then dose maintenance for 3 weeks; then downward titration of SPD503 at 1 mg weekly decrements for 3 weeks while maintaining the subject's current psychostimulant dose and frequency.
Groups:
- Methylphenidate + SPD503: Each group received SPD503 (Guanfacine hydrochloride) at doses up to 4 mg/day coadministered with the psychostimulant. Methylphenidate was dosed according to the prescribing physician's instructions.
- Amphetamine + SPD503: Each group received SPD503 (Guanfacine hydrochloride) at doses up to 4 mg/day coadministered with the psychostimulant. Amphetamine was dosed according to the prescribing physician's instructions.
Period: Overall Study
Arm/Group | Methylphenidate + SPD503 | Amphetamine + SPD503
Started | 42 | 33
Completed | 37 | 26
Not Completed | 5 | 7
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Sponsor's decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate + SPD503 | Amphetamine + SPD503 | Total
Number analyzed (Participants) | 42 | 33 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 33 | 75
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (1.79) | 11.6 (2.62) | 11.4 (2.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 29 | 26 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 33 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS-IV) Total Score at 6 Weeks
Description: Change in the Attention Deficit Hyperactivity Disorder Rating Scale-fourth edition (ADHD-RS-IV) total score from baseline. The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and 6 weeks
Population: Full Analysis Set (FAS) defined as all subjects with a baseline and at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Methylphenidate + SPD503 | Amphetamine + SPD503
Number analyzed (Participants) | 42 | 32
Units on a Scale | -17.8 (10.2) | -13.8 (11.19)
Statistical Analysis 1: Comparison: Methylphenidate + SPD503; Change from baseline in ADHD-RS-IV total score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Amphetamine + SPD503; Change from baseline in ADHD-RS-IV total score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 6 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Methylphenidate + SPD503 | Amphetamine + SPD503
Number analyzed (Participants) | 42 | 32
Participants | 28 | 18

3. Secondary Outcome: Change From Baseline in Conner's Parent Rating Scale-revised Short Version (CPRS-R) Total Score at 6 Weeks
Description: The Conner's Parent Rating Scale-revised short version (CPRS-R) consists of 27 questions graded on a scale from 0 (not true at all) to 3 (very much true) with a total score ranging from 0 to 81. Higher scores are indicative of increased ADHD. This scale allows parents to respond on the basis of the child's behavior and help assess ADHD and evaluate problem behavior.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Methylphenidate + SPD503 | Amphetamine + SPD503
Number analyzed (Participants) | 42 | 32
Units on a Scale | -22.18 (15.47) | -16.28 (18.12)
Statistical Analysis 1: Comparison: Methylphenidate + SPD503; Change from baseline in CPRS-R total score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Amphetamine + SPD503; Change from baseline in CPRS-R total score; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

4. Secondary Outcome: Number of Participants With Improvement on Parent Global Assessment (PGA) Scores
Description: Parent Global Assessment (PGA) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). The PGA is designed to capture parent's opinions of their child's disease (ADHD) severity and improvement. Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 6 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Methylphenidate + SPD503 | Amphetamine + SPD503
Number analyzed (Participants) | 42 | 32
Participants | 32 | 21

5. Secondary Outcome: Change From Baseline in Child Health Questionnaire-Parent Form (CHQ-PF50) Scores at 6 Weeks
Description: The Child Health Questionnaire-Parent Form (CHQ-PF50) was developed to measure the physical and psychosocial well-being of children aged 5 years of age and older. Total scoring ranges from 0-100 for each. Increases in scores represent improved well-being in subjects as assessed by their parents.
Time Frame: Baseline and 6 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Methylphenidate + SPD503 | Amphetamine + SPD503
Number analyzed (Participants) | 42 | 32
Units on a scale
  Physical Summary Score | -0.38 (5.83) | 0.22 (11.94)
  Psychosocial Summary Score | 8.98 (6.69) | 11.56 (10.00)
Statistical Analysis 1: Comparison: Methylphenidate + SPD503; Change in physical summary score; Test type: Superiority or Other; p = 0.7004, t-test, 2 sided
Statistical Analysis 2: Comparison: Methylphenidate + SPD503; Change in psychosocial summary score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Amphetamine + SPD503; Change in physical summary score; Test type: Superiority or Other; p = 0.9257, t-test, 2 sided
Statistical Analysis 4: Comparison: Amphetamine + SPD503; Change in psychosocial summary score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Methylphenidate + SPD503 | Amphetamine + SPD503
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/33
Other Adverse Events (participants affected / at risk) | 41/42 | 29/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate + SPD503 (N=42) | Amphetamine + SPD503 (N=33)
Abdominal pain upper (Gastrointestinal disorders) | 12 | 12
Constipation (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 15 | 11
Upper respiratory tract infection (Infections and infestations) | 6 | 2
Anorexia (Metabolism and nutrition disorders) | 3 | 3
Appetite increased (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 12 | 13
Sedation (Nervous system disorders) | 4 | 2
Somnolence (Nervous system disorders) | 6 | 8
Anxiety (Psychiatric disorders) | 6 | 5
Depressed mood (Psychiatric disorders) | 1 | 3
Initial insomnia (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 7 | 5
Irritability (Psychiatric disorders) | 10 | 14
Social avoidant behavior (Psychiatric disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.